CLINICAL TRIAL: NCT01911767
Title: Biogen Idec Multiple Sclerosis Pregnancy Exposure Registry
Brief Title: Biogen Multiple Sclerosis Pregnancy Exposure Registry
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS402
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis; Exposure During Pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate; peginterferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dimethyl fumarate: Exposure to dimethyl fumarate since the first day of her last menstrual period (LMP) prior to conception or at any time during pregnancy
  Interventions: Drug: Dimethyl fumarate
- Peginterferon beta-1a: Exposure to Peginterferon beta-1a since 17 days prior to the first day of her LMP prior to conception or at any time during pregnancy.
  Interventions: Drug: Peginterferon beta-1a
- Disease Modifying Therapy (DMT) Unexposed: Never received DMT therapy; discontinued treatment with any DMT at least more than 5× half-life prior to Day 1 of her LMP and throughout the entire pregnancy.

INTERVENTIONS:
Drug: Dimethyl fumarate — Administered as specified in treatment arm.
  Other Names: Tecfidera; BG00012; DMF
  Groups: Dimethyl fumarate
Drug: Peginterferon beta-1a — Administered as specified in treatment arm.
  Other Names: Plegridy; BIIB017
  Groups: Peginterferon beta-1a

SUMMARY:
The primary objective of the study is to prospectively evaluate pregnancy outcomes in women with multiple sclerosis who were exposed to a Registry-specified Biogen Multiple Sclerosis product during the eligibility window for that product. The Registry-specified Biogen MS products being studied are dimethyl fumarate, and Pegylated human interferon beta-1a. The secondary objective of the study is to prospectively evaluate pregnancy outcomes in women with MS who were unexposed to disease-modifying therapies (DMTs).

DETAILED DESCRIPTION:
The Biogen Multiple Sclerosis Pregnancy Exposure Registry is a prospective, observational registry designed to evaluate pregnancy outcomes in women with multiple sclerosis (MS) who were exposed to a Registry-specified Biogen Multiple Sclerosis product during the eligibility window for that product. Women of childbearing potential are a considerable segment of the patient population affected by MS and are likely to be exposed to a Registry-specified Biogen MS product around the time of conception and during pregnancy. Biogen completed pregnancy registries for Avonex and Tysabri; however, formal studies in pregnant women have not been conducted. Therefore, it is important to evaluate, in a global Pregnancy Registry, how exposure to a marketed Biogen MS product specified in this Pregnancy Registry may affect pregnancy and infant outcomes. Data will be collected on prospective pregnancies (i.e. enrollment prior to knowledge of outcome) at time of enrollment, 6 to 7 months gestation, and approximately 4,12, and 52 weeks after estimated date of delivery. The prevalence of spontaneous abortions, birth defects, and other pregnancy and infant outcomes will be calculated and compared to background rates from external sources such as the European Surveillance of Congenital Anomalies.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient consent
* Patient has a diagnosis of MS.
* Documentation that the patient was exposed to a Registry-specified Biogen MS product during the eligibility window for that product.
* DMF: Exposure since the first day of her last menstrual period (LMP) prior to conception or at any time during pregnancy.
* Peginterferon beta-1a: Exposure since 17 days prior to the first day of her LMP prior to conception or at any time during pregnancy.
* DMT unexposed pregnancy cohort: Never received DMT therapy
* Patient agrees to sign the Release of Medical Information Form, thereby permitting the Registry to contact her health care provider (HCP(s)) and the pediatric HCP for medical information.

Key Exclusion Criteria:

* The outcome of the pregnancy (i.e., pregnancy loss or live birth) must not be known at the time of enrollment.
* Initial maternal health assessment upon confirmation of pregnancy does not preclude participation in the Registry unless a patient tests positive for a medical condition associated with negative pregnancy outcomes (e.g., toxoplasmosis screen and syphilis [venereal disease research laboratory test and rapid plasma reagin test] blood screen) in the opinion of the healthcare provider (HCP).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Within each product cohort, approximately 310 to 375 pregnant women exposed to a Registry-specified Biogen MS product will be enrolled in order to observe 300 prospective pregnancy outcomes. The infants born to these women will also be part of the population studied. Patients with prenatal testing prior to enrollment (with the exception of a first trimester ultrasound to date the pregnancy) will not be counted towards the 300 prospective pregnancy outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy Loss | During pregnancy up to 52 weeks post-delivery
  * Elective or therapeutic pregnancy terminations (any induced or voluntary fetal loss during pregnancy)
  * Spontaneous abortions (<22 weeks of gestation)
  * Fetal death, including stillbirths (fetuses born dead at >=22 weeks of gestation), which will be further classified as follows:
  * early fetal loss (fetal death occurring at >=22 weeks but <28 weeks of gestation)
  * late fetal loss (occurring at >=28 weeks of gestation)
Live Birth | During pregnancy up to 52 Weeks Post-Delivery
  * Premature birth (delivered <37 weeks)
  * Full-term birth (delivered >=37 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- Research Site, Cambridge, Massachusetts, United States
- Research Site, Box Hill, Victoria, Australia
- Research Site, Cambridge, Massachusetts, Canada
- Research Site, Bron, Cedex, France
- Research Site, Bochum, Nordrhein Wesfalen, Germany
- Research Site, Dublin, Ireland
- Italy (5):
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Roma
- Research Site, Bialystok, Poland
- Spain (2):
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Salford, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Hellwig K, Rog D, McGuigan C, Houtchens MK, Bruen DR, Mokliatchouk O, Branco F, Peng X, Everage NJ. Interim Analysis of Pregnancy Outcomes After Exposure to Dimethyl Fumarate in a Prospective International Registry. Neurol Neuroimmunol Neuroinflamm. 2021 Nov 23;9(1):e1114. doi: 10.1212/NXI.0000000000001114. Print 2022 Jan. PMID 34815321